CLINICAL TRIAL: NCT06591169
Title: Polycystic Ovarian Syndrome Women with NAFLD and Obstructive Sleeping Apnea: Program of Lifestyle Changes
Brief Title: Lifestyle Changes in PCOS with OSA and NAFLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Giza, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005321
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: PCOS; NAFLD; OSA
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study (Experimental): this group will contain twenty obese females with a complaint of NAFLD, PCOS and OSA. for eight weeks, these obese females will receive metformin tablet (thrice daily), program of low diet intake, and daily walking for 30 minutes
  Interventions: Behavioral: diet restriction and exercise
- control group (Active Comparator): this group will contain twenty obese females with a complaint of NAFLD, PCOS and OSA. for eight weeks, these obese females will receive metformin tablet (thrice daily) and program of low diet intake
  Interventions: Behavioral: diet restriction

INTERVENTIONS:
Behavioral: diet restriction and exercise — this group will contain twenty obese females with a complaint of NAFLD, PCOS and OSA. for eight weeks, these obese females will receive metformin tablet (thrice daily), program of low diet intake, and daily walking for 30 minutes
  Arms: study
Behavioral: diet restriction — this group will contain twenty obese females with a complaint of NAFLD, PCOS and OSA. for eight weeks, these obese females will receive metformin tablet (thrice daily) and program of low diet intake
  Arms: control group

SUMMARY:
Complain of obstructive sleeping apnea and fatty liver is common in PCOS women so lifestyle changes are recommended

DETAILED DESCRIPTION:
Forty obese PCOS men with obstructive sleeping apnea and compaint of fatty liver will participate in this trial . Group (study group) will contain twenty obese females with a complaint of PCOS and OSA and fatty liver. for eight weeks, these obese females will receive metformin tablet (thrice daily), program of low diet intake, and daily walking for 30 minutes. Group (control group) will contain twenty obese females with a complaint of PCOS and OSA and fatty liver . for eight weeks, these obese females will receive metformin tablet (thrice daily), program of low diet intake,

ELIGIBILITY:
Inclusion Criteria:

* forty women
* women complaint PCOS
* women complain obstructive sleep apnea
* women are obese
* women complain fatty liver

Exclusion Criteria:

* cardiac insult
* renal insult
* malignacy
* pregnancy

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-identified national gender ID
Enrollment: 40 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
aspartate transamianse | it will be assessed in serum after eight weeks

SECONDARY OUTCOMES:
alanine transaminase | it will be assessed in serum after eight weeks
triglycerides | it will be assessed in serum after eight weeks
neck circumference | it will be assessed after eight weeks
waist circumference | it will be assessed after eight weeks
body mass index | it will be assessed after eight weeks
testesterone | it will be assessed in serum after eight weeks
ratio of luteinizing hormone and follicle-stimulating hormone | it will be assessed after eight weeks
apnea hyopnea index | it will be assessed after eight weeks
Epworth sleeping scale | it will be assessed after eight weeks
Dehydroepiandrosterone | it will be assessed in serum after eight weeks
waist hip ratio | it will be assessed after eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt